CLINICAL TRIAL: NCT03753113
Title: Evaluating the Efficacy of Topical Herbal Solution on the Treatment of Androgenetic Alopecia and Comparison With Minoxidil 5%: A Double-Blind, Randomized, Clinical Trial Study
Brief Title: Evaluating the Topical Herbal Solution on the Treatment of Male Pattern Hair Loss and Comparison With Minoxidil 5%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Farid Masoud (Other)
Responsible Party: Sponsor-Investigator, Farid Masoud, Principal Investigator, Tabriz University of Medical Sciences
Organization: Tabriz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TabrizUMS
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Androgenetic Alopecia
Keywords: Androgenic Alopecia; Hair Diseases; Skin Diseases; Baldness; Alopecia; Hair Loss
MeSH Terms: conditions — Alopecia; Hair Diseases; Skin Diseases | interventions — Minoxidil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): The patients will be applied 1 mL of solutions(Herbal and Minoxidil) at morning and evening intervals to the thinning hair areas of the scalp for 36 weeks.
  Interventions: Drug: Topical Herbal Solution; Drug: Topical Minoxidil 5%
- Control group (Active Comparator): The patients will be applied 1 mL of Minoxidil 5% solutions at morning and evening intervals to the thinning hair areas of the scalp for 36 weeks.
  Interventions: Drug: Topical Minoxidil 5%

INTERVENTIONS:
Drug: Topical Herbal Solution — Use Topical Herbal Solution every day in scalp hair loss areas for 36 weeks.
  Arms: Treatment group
Drug: Topical Minoxidil 5% — Use Minoxidil 5% solution every day in scalp hair loss areas for 36 weeks.
  Other Names: Minoxidil

SUMMARY:
The purpose of this study is evaluating the efficacy and safety of a topical herbal solution in males for the treatment of Androgenetic alopecia.

DETAILED DESCRIPTION:
This study will be done on male subjects with Androgenetic alopecia(AGA). The patients will be selected by volunteers attending the Dermatology department of Sina Hospital, and eligible individuals will be selected among them. Subjects were randomized to use either Topical Herbal Solution or Topical Minoxidil 5% for 36 weeks.

To our knowledge, this herbal solution for the first time covers all four major causes of AGA, including the 5α-reductase enzyme, androgen receptors, paracrine agents that affecting dermal papilla and hair cell apoptosis processes. Therefore it acts with the quadruple mechanism. The application of this new herbal solution for the treatment of AGA should be recommended.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 to 50 years old
* Written consent
* Normal general health status
* Men who have a presentation of androgenetic alopecia (Norwood II - V).

Exclusion Criteria:

* Use of any topical product in the target region interfering with the study product in the last three months
* Within the past 6 months receiving of chemotherapy/cytotoxic agents
* Clinical diagnosis of alopecia areata or other non-AGA forms of alopecia
* Uncontrolled hypertension
* Any dermatological disorders in the scalp, such as fungal or bacterial infections, eczema, atopic dermatitis, seborrheic dermatitis, psoriasis, sun damage, skin cancer
* Hormonal diseases such as thyroid disorders, diabetes and, ...
* Smokers
* Liver and kidney disease
* History of hair transplants
* History of surgical correction of hair loss on the scalp
* Subject having dyed, bleached hair or, with a permanent wave prior to study start.
* No written consent

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy men 18 to 50 years old
Enrollment: 24 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farid Masoud, PharmD, Principal Investigator — Pharmacy Faculty; Yousef Javadzadeh, Ph.D, Study Director — Department of Pharmaceutics, Pharmacy Faculty; Hamideh Azimi Alamdari, MD, Principal Investigator — Department of Dermatology, Faculty of Medicine; Solmaz Asnaashari, Ph.D, Study Director — Department of Pharmacognosy, Pharmacy Faculty; Javad Shokri, Ph.D, Study Director — Department of Pharmaceutics, Pharmacy Faculty
Locations (1):
- Department of Dermatology, Sina Hospital, Tabriz, East Azerbaijan Province, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masoud F, Alamdari HA, Asnaashari S, Shokri J, Javadzadeh Y. Efficacy and safety of a novel herbal solution for the treatment of androgenetic alopecia and comparison with 5% minoxidil: A double-blind, randomized controlled trial study. Dermatol Ther. 2020 Nov;33(6):e14467. doi: 10.1111/dth.14467. Epub 2020 Nov 5. PMID 33112463

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: The patients applied 1 mL of solutions at morning and evening intervals to the thinning hair areas of the scalp for 36 weeks.
  Topical Herbal Solution: Use Topical Herbal Solution every day in scalp hair loss areas for 36 weeks.
  Topical Minoxidil 5%: Use Minoxidil 5% solution every day in scalp hair loss areas for 36 weeks.
- Control Group: The patients applied 1 mL of solution at morning and evening intervals to the thinning hair areas of the scalp for 36 weeks.
  Topical Minoxidil 5%: Use Minoxidil 5% solution every day in scalp hair loss areas for 36 weeks.
Period: Overall Study
Arm/Group | Treatment Group | Control Group
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: At the Week 0 administration, subject demographics, hair diameter, and duration of androgenetic alopecia acquired.
Groups:
- Control Group: The patients applied 1 mL of solution at morning and evening intervals to the thinning hair areas of the scalp for 36 weeks
  Topical Minoxidil 5%: Use Minoxidil 5% solution every day in scalp hair loss areas for 36 weeks.
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Control Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.45 (5.744) | 33.67 (6.065) | 33.04 (5.812)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  Iran | 12 | 12 | 24
Hair diameter [Mean (Standard Deviation); unit: micrometer] | 52.75 (8.74) | 54 (6.729) | 53.38 (7.65)
Duration of androgenetic alopecia [Mean (Standard Deviation); unit: years] | 4.58 (2.24) | 4.42 (2.47) | 4.5 (2.3)
Family history of androgenetic alopecia [Count of Participants; unit: Participants]
  Yes | 10 | 9 | 19
  No | 2 | 3 | 5
Family history of the disease [Count of Participants; unit: Participants]
  Hypo/Hyperthyroidism | 5 | 3 | 8
  Cardiovascular | 2 | 2 | 4
  Diabetes | 1 | 1 | 2
  None | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Hair Diameter
Description: Change in hair diameter over time as compared to Baseline. Hair diameter measured via a digital micrometer.
Time Frame: baseline, 12, 24, and 36 weeks
Measure: Mean (Standard Deviation); unit: micrometer
Groups:
- Treatment Group: The patients applied 1 mL of solutions at morning and evening intervals to the thinning hair areas of the scalp for 36 weeks
  Topical Herbal Solution: Use Topical Herbal Solution every day in scalp hair loss areas for 9 months
  Topical Minoxidil 5%: Use Minoxidil 5% solution every day in scalp hair loss areas for 9 months
- Control Group: The patients applied 1 mL of solution at morning and evening intervals to the thinning hair areas of the scalp for 36 weeks
  Topical Minoxidil 5%: Use Minoxidil 5% solution every day in scalp hair loss areas for 9 months
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 12
micrometer
  Week 12 | 57.42 (8.88) | 51.58 (7.67)
  Week 24 | 60.92 (7.35) | 51.17 (7.82)
  Week 36 | 62.67 (7.19) | 50.58 (7.38)

2. Secondary Outcome: Patients Self - Assessment Questionnaire
Description: Self-administered hair growth questionnaire, consisting of 4 questions in the patient's language on treatment efficacy and three questions on satisfaction with appearance. For differences between self-assessment questionnaires. This questionnaire following 5-point scale: 1 = very satisfied, 2 = satisfied, 3 = neutral (neither satisfied nor dissatisfied), 4 = dissatisfied, 5 = very dissatisfied. Higher scores indicated a worse outcome.
Time Frame: through study completion
Population: All participants for whom data were collected at weeks 36.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 12
score on a scale | 1.25 (0.452) | 2.58 (0.669)

3. Secondary Outcome: Adverse Events
Description: Incidence of adverse events such as itching, redness, inflammation etc
Time Frame: baseline, 12, 24, and 36 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group | Control Group
Number analyzed (Participants) | 12 | 12
Participants
  scalp itching | 1 | 4
  scalp dryness | 0 | 2
  headache | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the beginning of the study until 9 months
Description: According to its herbal origin and topical administration, In both groups, neither all-cause mortality nor serious adverse events were reported.
Arm/Group | Treatment Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=12) | Control Group (N=12)
Blurred vision (Eye disorders) | 0 | 0
Chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=12) | Control Group (N=12)
scalp itching (Skin and subcutaneous tissue disorders) | 1 | 4
scalp dryness (Skin and subcutaneous tissue disorders) | 0 | 2
headache (Nervous system disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
Small numbers of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-08-08): https://cdn.clinicaltrials.gov/large-docs/13/NCT03753113/Prot_SAP_ICF_000.pdf